CLINICAL TRIAL: NCT05339113
Title: Comparison of [68Ga]GaFAPI-46 PET/CT and [18F]FDG PET/CT Findings in Breast Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The National Center of Oncology, Azerbaijan (Other Government)
Collaborators: SOFIE INC (Unknown)
Responsible Party: Principal Investigator, Fuad Novruzov, Head of Nuclear Medicine Department, The National Center of Oncology, Azerbaijan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCO-21001
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Breast Neoplasms; Positron Emission Tomography; Fibroblast Activation Protein Inhibitor; Fluorodeoxyglucose F18
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-46 PET/CT + 18-FDG PET/CT (Experimental): 18FDG PET/CT scan is followed by [68Ga]FAPI-46 PET/CT within 2-3 days.
  Interventions: Diagnostic Test: 68Ga-FAPI-46 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 PET/CT — Patients are scanned 10 minute, 30 minute and 1 hour after 68Ga-FAPI-46 as well as one hour 18-FDG injection within 2-3 days interval.

SUMMARY:
The aim of this study is to compare the diagnostic performance of 68Ga-FAPI-46 PET/CT and 18F-FDG PET/CT in primary and metastatic lesions of breast cancer and to reveal the best diagnostic imaging time of 68Ga-FAPI-46 PET/CT.

DETAILED DESCRIPTION:
Participants with breast carcinoma will undergo contemporaneous 18F-FDG and 68Ga-FAPI PET/CT. Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 68Ga-FAPI PET/CT will be calculated and compared to evaluate the diagnostic efficacy. In addition, best diagnostic imaging time of 68Ga-FAPI-46 PET/CT will be evaluated at 10th, 30th and 60th minute scan time.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (aged 18 years or order);
* participants with newly diagnosed breast carcinoma;
* pathology confirmed by lesion tru-cut biopsy;
* participants who were able to provide informed consent.

Exclusion Criteria:

* participants with non-malignant lesions;
* participants with pregnancy;
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum standardised uptake value [SUVmax] for primary lesion | 2-3 days
  SUVmax of 68Ga-FAPI PET/CT for breast carcinoma in comparison with SUVmax value of 18F-FDG PET/CT
Best diagnostic imaging time of 68GaFAPI-46 PET/CT | 2-3 days
  Tumor-to-background ratio values measured over the 10th, 30th and 60th minute scan time

SECONDARY OUTCOMES:
Diagnostic efficacy for breast carcinomas | 2 days
  Sensitivity, specificity, accuracy, positive predictive value (PPV) and negative predictive value (NPV) of 68Ga-FAPI PET/CT for breast carcinomas in comparison with 18F-FDG PET/CT
SUVmax for metastatic lymph nodes | 2 days
  SUVmax of 68Ga-FAPI PET/CT for metastatic lymph nodes in comparison with 18F-FDG PET/CT
Diagnostic efficacy for metastatic lymph nodes | 2 days
  Sensitivity, specificity, accuracy, PPV and NPV of 68Ga-FAPI PET/CT for metastatic lymph nodes in comparison with 18F-FDG PET/CT
Correlation between tumor SUVmax values and pathology grade | 2 days
  Correlation between tumor SUVmax values and pathology grade calculated

CONTACTS AND LOCATIONS:
Locations (1):
- National Centre of Oncology, Baku, Azerbaijan